CLINICAL TRIAL: NCT06441552
Title: Learning the Natural History of Recovery After Stroke - Cognitive, Motor and Sensory Function
Brief Title: The Natural History of Recovery After Stroke
Acronym: RESTRO
Status: Recruiting | Type: Observational
Sponsor: Adi Negev-Nahalat Eran (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: ADINEGEV-2023_106; SIS70023GR0026 (Other Grant/Funding Number: KB6NZDMMP3N8)
Record Dates: First submitted 2024-04-30; First posted 2024-06-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Vascular Accident (CVA)/Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ofakim: Non-interventional group, recruited at Adi-Negev Rehabilitation Center, Israel.
  Interventions: Other: non-interventional
- Haifa: Non-interventional group, recruited at Rambam Health Care Campus, Israel.
  Interventions: Other: non-interventional
- Hebron: Non-interventional group, recruited through Green Land Society for Health Development, Palestine.
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
The goal of this longitudinal observational study is to learn the course of recovery after stroke. Specifically, in this study we will learn and describe the changes in cognitive, motor and sensory function over time in stroke patients.

DETAILED DESCRIPTION:
This study constitutes the first step in the RESTRO project: Evaluation of an accessible and affordable neurorehabilitation program to promote recovery and to enhance the quality of life after stroke. In this study, we will monitor sensorimotor and cognitive functions of Stroke patients along the first 6 to 12 month following their stroke. Data from three primary sites will be collected and compared in several time points, and its relation to the type and intensity of the rehabilitation program, usually provided in each site, will be tested.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Independent in all activities of daily living before the stroke.
* In- and out-patients at Adi-Negev Nahalat-Eran rehabilitation center, with first ever stroke, or with a recurrent stroke that did not lead to disability (were independent in ADL before the second stroke).
* Medically stable
* Able to provide informed consent.

Exclusion Criteria:

* The presence of any degenerative neurological condition, neuropathy, myopathy or Polio that are not secondary to stroke, excluding diabetic related changes.
* Traumatic brain injury and/or extra-cerebral hemorrhage.
* Significant psychiatric condition, including alcoholism and drug abuse.
* Any severe orthopedic condition (such as amputation or severe pain that limits activity) or chronic pain syndrome.
* Participation in another interventional study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke survivors and healthy adults.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Fugl-Meyer Assessment:
  Motor score is on a 0-100 scale. High score is better.
Action Research Arm Test (ARAT) | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Action Research Arm Test Score is on a 0-57 scale. High score is better.
10-meter walk test (10MWT) | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Outcome is the average walking velocity over 10 meters. Measured in m/sec.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | Baseline (<3weeks)
  measure of stroke severity on a 0-42 scale, with lower scores indicates lower severity (lower is better).
The Stroke Self-Efficacy Questionnaire (SSEQ) | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  This is a self-reported ability perception scale. Outcome range is 0-130 with higher scores indicate a better self-perceived ability.
The Nine Hole Peg Test (NHPT) | Baseline (<3weeks), 1-year
  This is an upper extremity dexterity test. Outcome is the time taken to complete the task. Measured in sec.
The Functional Dexterity Test (FDT) | Baseline (<3weeks), 1-year
  This is an upper extremity dexterity test. Outcome is the time taken to complete the task. Measured in sec.
The Behavioral Inattention Test (BIT) | Baseline (<3weeks)
  This is an instrument aimed at detecting visual neglect. In this study we use only two subsections of the test: star cancellation (scored on a 0-54 scale) and representational drawing (scored on a 0-3 scale). For both, higher scores are better.
The Ashworth scale | Baseline (<3weeks)
  This instrument is used to detect spasticity (increased muscle tone). Outcome is 0-4 scale, with lower scores means better outcome (less spasticity).
Kinetics-fingers1 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  To measure fingers kinetics, we will use a custom-built device that measures finger force for flexion and extension. Outcome is the force in Newtons (N) generated by each finger.
Kinetics-fingers2 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  To measure fingers kinetics, we will use a custom-built device that measures finger force for flexion and extension. Outcome measure is the Individuation Index, measured in arbitrary units (a.u.). The individuation index is calculated as the ratio between the forces generated by the non-instructed digits and the force generated by the instructed digit. This index evaluates the ability to generate force in each digit independently of the other digits.
Kinetics-grip | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Grip force will be measured using the microFET Digital HandGrip Dynamometer (Hoggan Scientific). Outcome is the maximal force in Newtons.
Kinematics-reaching | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Kinematic measurements of upper extremity reaching task:
  Kinematic measures will be extracted using markerless pose estimation algorithms (such as OpenPose and MediaPipe). Reaching error (distance of the hand from the target) and reaching extent (maximum distance of the wriest from the shoulder). Measured in mm.
Kinematics-duration | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Kinematic measurements of upper extremity reaching tasks:
  Kinematic measures will be extracted using markerless pose estimation algorithms (such as OpenPose and MediaPipe). Reaching duration. Measured in seconds.
Kinematics-smoothness | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Kinematic measurements of upper extremity reaching tasks:
  Kinematic measures will be extracted using markerless pose estimation algorithms (such as OpenPose and MediaPipe). Reaching smoothness as the integrated jerk (as described by Platz et al. 1994, Dimensions are L^2/T^6) and the spectral arch length (as described by Balasubramanian et al. 2015).
Kinematics-Inter-joint coordination | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Kinematic measurements of upper extremity reaching tasks:
  Kinematic measures will be extracted using markerless pose estimation algorithms (such as OpenPose and MediaPipe). Inter-joint coordination will be measured through computing the cross correlation between elbow, writs and shoulder joint angles and the proportion of time when joints flexed or extend together. Arbitrary units.
Rehabilitation-intensity | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Number of rehabilitative sessions per week, in total and for each modality separately (e.g., physical therapy, occupational therapy, etc.)
Rehabilitation-time | one or more of: Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Time, in minutes, of each therapy session.
Rehabilitation-period | one or more of: Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Period of time (in month) for which the participant received therapy.
Supporting data-age | Baseline
  Age at admission, in years.
Supporting data-sex | Baseline
  Biological Male or Female
Supporting data-time1 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  time from stroke onset in days
Supporting data-time2 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  other time periods (e.g., inpatient time, rehabilitation duration, etc.) in Months.
anthropometric data-height | Baseline
  Height in cm
anthropometric data-weight | Baseline
  Weight in kg
supporting data-directional | Baseline
  affected brain side: L/R/Both affected body side: L/R/Both hand dominance: L/R leg dominance: L/R
supporting data-medical history | Baseline
  Any relevant history of illnesses.
Cognition-impairment | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Montreal Cognitive Assessment (MoCA). 0-30 scale with higher values indicate better cognitive state.
Cognition-inhibition1 | one or more of : Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Percent correct responses in an anti-saccade computerized task.
Cognition-inhibition2 | one or more of : Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Reaction time (in msec) in an anti-saccade computerized task.
Timed up and Go test (TUG) | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Time taken to complete the TUG task. Measured in seconds.
Gait Specific attentional profile (G-SAP) | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  This is a questioner aimed at evaluating the attentional profile of the patient during walking. It has several subscales measured on a Likert 5-point scale. Total score range is 11-55 with lower values indicate better outcome.
Gait analysis-temporal | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gait analysis while participants are walking on a treadmill (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany) with an embedded force sensors array. Temporal measures include step and stride time. Measured in seconds.
Gait analysis-spatial | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gait analysis while participants are walking on a treadmill (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany) with an embedded force sensors array. Spatial measures include step and stride length and width. Measured in meters.
Gait analysis-steadiness | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gait analysis while participants are walking on a treadmill (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany) with an embedded force sensors array. Steadiness is measured by calculating the maximal Lyapunov exponent of the center of pressure dynamics (as described by Rosenstein et al. 1993). Units of measure are arbitrary.
Gaze-angle1 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gaze behavior during walking using a mobile eye-tracker (Pupil Invisible, Pupil Labs, Germany). Head, eye and gaze (head and eye combined) angles on the sagittal and horizontal planes will be measured. Outcome in degrees.
Gaze-angle2 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gaze behavior during walking using a mobile eye-tracker (Pupil Invisible, Pupil Labs, Germany). Gaze angles will be measured relative to the vanishing point. Outcome in %.
Gaze-downward | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gaze behavior during walking using a mobile eye-tracker (Pupil Invisible, Pupil Labs, Germany). Time spent looking onto the walking surface. Outcome in %.
Gaze-look-ahead distance | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Gaze behavior during walking using a mobile eye-tracker (Pupil Invisible, Pupil Labs, Germany). Look-ahead distance. Outcome in meters.
Balance-Berg | baseline
  Berg Balance Scale (BBS) measured on a 0-56 scale with higher score represent better outcome.
Balance-postural steadiness1 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Postural Sway (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany). Outcome is sway range in mm.
Balance-postural steadiness2 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Postural Sway (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany). Outcome is sway velocity in mm/sec.
Balance-postural steadiness3 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Postural Sway (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany). Outcome is sway area in mm^2.
Balance-postural steadiness4 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Postural Sway (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany). Outcome is the short-term diffusion coefficients, as described by Collins and De-Luka (1993), measured in mm^2/sec.
Habitual activity1 | one or more of :Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Monitoring habitual activity during hospital stay. Time spent walking, sitting and laying in hours/day. Measured over 3-5 consecutive days.
Habitual activity2 | one or more of :Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Monitoring habitual activity during hospital stay. Distance walked in meters/day. Measured over 3-5 consecutive days.
Sensory-tactile | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Sensory acuity will be measured using Semmes-Weinstein monofilament. Outcome is in grams.
Coordination-LE1 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  LEMOCOT- Lower Extremity Motor Coordinating Test. Outcome is the number of touches (count).
Coordination-LE2 | Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  LEMOCOT- Lower Extremity Motor Coordinating Test. Outcome is the touches' errors (distance from the middle of the target), measured in mm. To measure errors, the LEMOCOT will be performed on an array of force sensors (Zebris FDM-T Treadmill, Zebris Medical GmbH, Germany) that detects the touches position.
Reticulospinal excitability | one or more of: Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  Response enhancement following a startling auditory stimuli (StartReact measure). Reaction time is measured in msec based on EMG signal from the wrist extensors and biceps (gtech USB-Amp). The StartReact measure is the enhancement in reaction time in the startle condition (LED+105Db auditory stimulus) compared to a control condition (LED+80Db auditory stimulus)
Muscle controllability1 | one or more of: Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  The ability to control a cursor in a virtual environment using EMG recordings from wrist extensors and biceps (Trigno Wireless EMG System, Delsys, USA). Outcome is success rate in %.
Muscle controllability2 | one or more of: Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  The ability to control a cursor in a virtual environment using EMG recordings from wrist extensors and biceps (Trigno Wireless EMG System, Delsys, USA). Outcome is time to target sec.
Muscle controllability3 | one or more of: Baseline (<3weeks), 1-month, 3-month, 6-month, 1-year
  The ability to control a cursor in a virtual environment using EMG recordings from wrist extensors and biceps (Trigno Wireless EMG System, Delsys, USA). Outcome is path length in cm.
Neuroimaging | one or more of :1-month, 3-month, 6-month, 1-year
  CT/MRI based structural neuroimaging. Outcomes are the areas affected by stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bar-Haim, PhD, Principal Investigator — Ben-Gurion University of the Negev; Lior Smuelof, PhD, Principal Investigator — Ben-Gurion University of the Negev; Shirley Handelzalts, PhD, Principal Investigator — Ben-Gurion University of the Negev; Firas Mawase, PhD, Principal Investigator — Technion, Israel Institute of Technology; Akram Amro, PhD, Principal Investigator — Green Land Society for Health Development
Locations (3):
- Israel (2):
  - Rambam/Technion, Haifa
  - Adi-Negev Nahalat Eran, Ofakim
- Al-Ahli hospital, Hebron, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Background] Rosenstein, M. T., Collins, J. J., & De Luca, C. J. (1993). A practical method for calculating largest Lyapunov exponents from small data sets. Physica D: Nonlinear Phenomena, 65(1-2), 117-134.
- [Background] Platz T, Denzler P, Kaden B, Mauritz KH. Motor learning after recovery from hemiparesis. Neuropsychologia. 1994 Oct;32(10):1209-23. doi: 10.1016/0028-3932(94)90103-1. PMID 7845561
- [Background] Balasubramanian S, Melendez-Calderon A, Roby-Brami A, Burdet E. On the analysis of movement smoothness. J Neuroeng Rehabil. 2015 Dec 9;12:112. doi: 10.1186/s12984-015-0090-9. PMID 26651329
- [Background] Collins JJ, De Luca CJ. Open-loop and closed-loop control of posture: a random-walk analysis of center-of-pressure trajectories. Exp Brain Res. 1993;95(2):308-18. doi: 10.1007/BF00229788. PMID 8224055